CLINICAL TRIAL: NCT02013115
Title: Curosurf/Budesonide for Infants With Respiratory Distress Syndrome
Acronym: Budesonide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Chen Long,MD, MD, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: curosurf/Budesonide for NRDS
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2013-12

CONDITIONS: Respiratory Distress Syndrome
Keywords: infant; respiratory distress syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cursurf (No Intervention): The baby with respiratory distress syndrome was given Cursurf through intubation.
- Cursurf and Budesonide (Experimental): The baby with respiratory distress syndrome was given Cursurf and Budesonide through intubation.
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: Budesonide — Experimental: Cursurf and Budesonide The baby with respiratory distress syndrome was given Cursurf and Budesonide through intubation
  Other Names: Pumicort
  Arms: Cursurf and Budesonide

SUMMARY:
Infants showing high local pulmonary inflammation diagnosted by respiratory distress syndrome usually need the second or more pulmonary surfactant and is easier to developing to Brochopulmonary. Cursurf is used worldwide in infants with respiratory distress syndrome, Budesonide is a glucocorticoid with a high local anti-inflammatory effect.Our hypothesis is Cursurf combined with Budesonide could reduced the need of Cursurf and incidence of Brochopulmonary dysplasia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of respiratory distress syndrome

Exclusion Criteria:

* pneumothorax
* surgical disease
* major congenical defects

Max Age: 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
need of pulmonary surfactant | one month
  The hypothesis is Cursurf/Budesonide could reduced the need of pulmonary surfactant

SECONDARY OUTCOMES:
the incidence of bronchopulmonary dysplasia | gestional age 36 weeks or later
  the hypothesis is Cursurf and Budesonide could reduced the incidence of bronchopulmonary dysplasia.

OTHER OUTCOMES:
need of intubation | one month
  The hypothesis is Cursurf/Budesonide could reduced the need of intubation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics, Daping Hospital, Research Institute of Surgery, Third Military Medical University, Chongqing, Chongqing Municipality, China